CLINICAL TRIAL: NCT05010135
Title: Evaluation of Balance and Gait Weight Distribution in Patients With Vertebral Column Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Dr. Anthony Kwok, Associate Professor, Tung Wah College
Other Study IDs: TungWC
Record Dates: First submitted 2021-02-18; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Vertebral Fracture; Balance; Gait, Unsteady
Keywords: Vertebral fracture; Balance; Gait
MeSH Terms: conditions — Spinal Fractures; Gait Disorders, Neurologic | interventions — Hand Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subject: Aged 60 and over. Male or Female. Able to give consent, and attend the assessment centre for the balance and gait weight distribution assessment.
  Interventions: Device: Zebris Gait System assessment for gait weight distribution + EMG evaluation of Quadriceps, Hamstrings, Tib Anterior and Calves + Positional Sense assessment
- Vertebral fracture subjects: Aged 60 or over. Male or Female. Able to give consent, and attend the assessment centre for the balance and gait weight distribution assessment.
  Have been diagnosed by doctors to have the vertebral fracture
  Interventions: Device: Zebris Gait System assessment for gait weight distribution + EMG evaluation of Quadriceps, Hamstrings, Tib Anterior and Calves + Positional Sense assessment

INTERVENTIONS:
Device: Zebris Gait System assessment for gait weight distribution + EMG evaluation of Quadriceps, Hamstrings, Tib Anterior and Calves + Positional Sense assessment — To measure the above parameters and to compare between the healthy subjects and the vertebral fracture subjects
  Other Names: TechnoBody Balance assessment: open eyes, closed eyes, single stand and double legs stand; Humac Norm assessment for the Quadriceps and Hamstring strength; Numeric Pain Rating Scale; Roland-Morris Disability Questionnaire; Oswestry Disability Index, SF-12, 6-meters Up and Go test; Hand Grip Strength, Fexibility measurement

SUMMARY:
Vertebral column fracture presents a significant warning of subsequent osteoporotic fracture and frequent falls. The presence of an osteoporotic vertebral fracture is also a predictor of further risk of vertebral and other osteoporotic fractures. This study provides balance assessment and gait evaluation for subjects with a known vertebral fracture.

Subjects are the known cases of vertebral fracture living in the community. They will be assessed for their balance and gait weight distribution by the TechnoBody for their balance ability, and the Zebris Gait System for the gait weight distribution. The Humac Norm for the lower limb muscle strength.

DETAILED DESCRIPTION:
This study evaluates the balance and weight distribution in walking gait in subjects with vertebral column fracture, comparing with the healthy subjects.

Study Objectives:

1. To evaluate the balance and gait weight distribution of the vertebral fracture patients.
2. To analyze the association between balance and gait weight distribution with fall risks in patients with stable vertebral fractures.
3. To construct a community fall prevention protocol.

Methodology:

Subjects:80 ambulatory subjects with a history of vertebral fracture, aged 60 and above, will be recruited from the community.

Study Design: an observational study by convenient sampling design.

Sample size calculation:

The calculated sample size of vertebral column fractures is 64. Allowing a 20% dropout rate, the round-up figure is 80.

Assessments will include the following:

1. . A questionnaire to collect the following information: i. Subjects' demographics, medical and medication history, and fall history. ii. Numeric Pain Rating Scale; ii. Roland-Morris Disability Questionnaire; iii. Oswestry Disability Index (Chinese version); iv. SF-12;
2. A 6-meters Up and Go test;
3. Hand Grip Strength to evaluate the muscle strength of the subjects
4. Flexibility measurement (how far to lean forward);
5. Balance and Centre of Gravity evaluation by the TechnoBody Machine;
6. . Zebris Gait System for their gait weight distribution evaluation, and
7. Humac Norm for the Quadriceps and Hamstrings muscle strength (both sides).

Statistical Analysis:

1. Statistical analyses will be performed using SPSS (version 24).
2. Two-sided tests and an α-level of 5% were used as the level of significance.
3. Chi-square tests were used for categorical variables.
4. Two-sample independent t-tests were used for continuous variables.

The balance, gait weight distribution pattern, and muscle strength will be analyzed by ANOVA.

Correlation analysis will be conducted for the factors of gender, age, and comorbid conditions.

From the results, strategies for fall prevention will be modelled and formulated.

Inclusion Criteria:

1. All subjects are aged 60 or above with a history of vertebral fracture, and able to walk without assistance;
2. Not received a bilateral hip replacement and spinal surgery;
3. No known malignance at time of enrollment;
4. Able to attend Tung Wah College for examination and assessment, understand, and sign the consent form.

Exclusion criteria:

1. Unable to attend the research center for receiving examination and tests;
2. Unable to give consent;
3. Diseases such as stroke and Parkinson's Disease that adversely affect the balance and gait weight distribution;
4. Bed-bound or wheel-chair bound patients.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects are aged 60 or above with a history of vertebral fracture, and able to walk without assistance;
2. Not received bilateral hip replacement and spinal surgery;
3. No known malignance at time of enrollment;
4. Able to attend Tung Wah College for examination and assessment, understand and sign the consent form.

Exclusion Criteria:

1. Unable to attend the research center for receiving examination and tests;
2. Unable to give consent;
3. Diseases such as stroke and Parkinson's Disease that adversely affect the balance and gait weight distribution;
4. Bed bound or wheel-chair bound patients.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All subjects are aged 60 or above with a history of vertebral fracture, and able to walk without assistance for vertebral fracture subjects.
  All subjects are aged 60 or above with no history of vertebral fracture, and able to walk without assistance for the healthy subjects.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Balance (measure by the TechnoBody machine to show the amplitude of body displacement from the centre) | Up to 24 weeks
  compare between the 2 groups
Gait weight distribution (measure by the Zebris Rehabwalk machine to show the force in Newton) | Up to 24 weeks
  compare between the 2 groups

SECONDARY OUTCOMES:
Muscle strength (measure by the Humac Norm machine to evaluate the Quadriceps and Hamstrings strength in Peak Torque, N) | Up to 24 weeks
  Compare between the 2 groups
Positional senses (measure by the position sensor attached on the feet, legs, thighs, lumber spine, thoracic spine and the cervical spine to show the body displacement in angle degrees). | Up to 24 weeks
  Compare between the 2 groups
Low Back Pain (measure by the Oswestry Disability Index and Roland Morris Disability Questionnaire) | Up to 24 weeks
  Compare between the 2 groups
Quality of Life evaluation (measure by the SF-12 questionnaire) | Up to 24 weeks
  Compare between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Anthony WL Kwok, Ph.D, Principal Investigator — Tung Wah College
Locations (1):
- Anthony Kwok, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05010135/Prot_SAP_ICF_000.pdf